CLINICAL TRIAL: NCT03352687
Title: Diaphragmatic Paralysis After Ultrasound Block of the Suprascapular Nerve for Shoulder Surgery : Incidence and Influence of the Approach
Brief Title: Diaphragmatic Paralysis After Ultrasound Block of the Suprascapular Nerve for Shoulder Surgery
Acronym: SSParaDia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0141; 2017-A01378-45 (Registry Identifier: ANSM register)
Record Dates: First submitted 2017-11-14; First posted 2017-11-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2019-04

CONDITIONS: Surgery
Keywords: Shoulder surgery; Local regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior SSAX (Experimental): patients receiving suprascapular and axillary nerve block (SSAX) whose approach to the SS nerve is performed by anterior route
  Interventions: Procedure: anterior SSAX
- Posterior SSAX (Experimental): patients receiving suprascapular and axillary nerve block (SSAX) whose approach to the SS nerve is performed by posterior route
  Interventions: Procedure: posterior SSAX

INTERVENTIONS:
Procedure: anterior SSAX — block of the suprascapular nerve block for shoulder surgery by anterior way
  Arms: Anterior SSAX
Procedure: posterior SSAX — block of the suprascapular nerve block for shoulder surgery by posterior way
  Arms: Posterior SSAX

SUMMARY:
Shoulder surgery is a source of intense postoperative pain that justifies the use of opioids. In this context, analgesia provided by locoregional anesthesia (ALR) improves the rehabilitation of patients by reducing the length of hospital stay and morphine consumption. Thus anesthesia of the brachial plexus interscalene (interscalene block or BIS) is considered as the reference technique for the management of post-operative pain after shoulder surgery. It is however provider of hemi-diaphragmatic paralysis (PhD) in nearly 100% of cases. Thus, this technique is usually avoided in patients with respiratory insufficiency. In arthroscopic shoulder surgery, the development of a suprascapular and axillary nerve (SSAX) conjugate block appears to be an effective analgesic alternative in this context.

DETAILED DESCRIPTION:
Two ultrasound-guided approaches of the suprascapular nerve (anterior and posterior approaches) have been described in the literature. From an anatomical point of view, the anterior approach could expose patients to the risk of ipsilateral PhD by phrenic nerve block secondary to diffusion of the local anesthetic into the supraclavicular region.

By measuring the diaphragm excursion during a sniff test, ultrasound allows reliable and reproducible analysis of the diaphragm function.

No study has evaluated the incidence of PhD after ultrasound block of the suprascapular nerve. Knowing the influence of the approach on this complication could be of major interest in this context.

ELIGIBILITY:
Inclusion Criteria:

* to benefit from scheduled arthroscopic surgery of the shoulder under general anesthesia
* Affiliate or beneficiary of a social security scheme
* Having signed the informed consent

Exclusion Criteria:

* the existence of contralateral diaphragmatic paralysis
* pre-existing respiratory insufficiency
* impossibility of performing diaphragmatic ultrasound
* the patient's refusal
* the existence of major spontaneous or acquired haemostatic disorders
* an infection at the point of puncture
* allergy to local anesthetics
* Pregnant or likely to be pregnant
* Patients under protection of the adults (guardianship, curators or safeguard of justice)
* Patients whose cognitive state does not allow assessment by the scales used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
change in diaphragmatic excursion | 30 minutes
  measured on ultrasound between the 30th minute after SSAX and the basal state (i.e. prior to regional anesthesia).
  The diaphragmatic excursion is the distance traveled by the diaphragm between the functional residual capacity (CRF) and the forced inspiration during a rapid voluntary sniffing (or "sniff test").

SECONDARY OUTCOMES:
PhD over time | Baseline, 30 minutes, 4 hours and 8 hours
  diaphragmatic excursion by a repeated ultrasound during a "sniff test" in the basal state (ie before regional anesthesia), then 30 minutes, 4 hours and finally 8 hours after realization of the ALR

OTHER OUTCOMES:
Pain evaluation by ENS | Baseline, 4 hours and 24 hours
  Evaluation of the pain by simple numerical scale (ENS from 0 to 10) in the post-interventional surveillance room (SSPI, at the 4th hour) and at the 24th hour
Morphine consumption | until 24 hours
  Evaluation of the morphine consumption in the post-interventional surveillance room (during 24 hours after the SSP)
patient's satisfaction | 24 hours
  Evaluation of the patient's satisfaction with the French Evaluation du Vécu de l'Anesthésie LocoRégionale (EVAN-LR) score

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice FERRE, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferre F, Pommier M, Laumonerie P, Ferrier A, Menut R, Bosch L, Balech V, Bonnevialle N, Minville V. Hemidiaphragmatic paralysis following ultrasound-guided anterior vs. posterior suprascapular nerve block: a double-blind, randomised control trial. Anaesthesia. 2020 Apr;75(4):499-508. doi: 10.1111/anae.14978. Epub 2020 Jan 26. PMID 31984478